CLINICAL TRIAL: NCT05468619
Title: A Phase I Adaptive, Multiple Dose Pharmacokinetic and Safety Assessment of Valacyclovir in Infants at Risk of Acquiring Neonatal Herpes Simplex Virus Disease
Brief Title: Neonatal Phase 1 Valacyclovir Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-0033; 5U54AI150225-05 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2022-07-21

CONDITIONS: Herpes Simplex
Keywords: Disease; Herpes Simplex Virus; Neonatal; Phase I; Valacyclovir
MeSH Terms: conditions — Herpes Simplex; Disease | interventions — Valacyclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): A cohort of neonates who are at risk of acquiring neonatal herpes simplex virus disease will receive 10 mg/kg of valacyclovir will be administered orally two times daily for 5 days. N=8
  Interventions: Drug: Valacyclovir
- Cohort 2 (Experimental): If the safety profile and the drug exposure concentrations in Cohort 1 are acceptable, eight new subjects will be enrolled in Cohort 2. If the mean of observed acyclovir exposures of subjects in Cohort 1 are below 24,000 ngxhr/mL, AND if no Grade 3 or Grade 4 AEs or SAEs are detected in any of the study subjects, then the 8 subjects enrolled in Cohort 2 will receive oral valacyclovir at a dose of 20 mg/kg administered two times daily for 5 days. Alternatively, if the mean of observed acyclovir exposures of subjects in Cohort 1 are above 48,000 ngxhr/mL AND if no Grade 3 or Grade 4 AEs or SAEs are detected in any of the study subjects, then the 8 subjects enrolled in Cohort 2 will receive oral valacyclovir at a dose that has been linearly adjusted downward to target 36,000 ngxh/mL area-under-the-concentration-time curve from 0 to 12 hours (AUC12).
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir is a L-valyl ester of acyclovir.

SUMMARY:
A Phase 1 study that will determine the valacyclovir dose that results in a systemic acyclovir exposure comparable to 10 mg/kg of parenterally administered acyclovir, which is an AUC0-12 of 24,000 ngxhr/mL to 48,000 ngxhr/mL. Neonates at risk of acquiring neonatal HSV will be enrolled in one of 2 cohorts. Cohort 1 will be comprised of eight subjects who will receive an initial dose of 10ml/kg of oral valacyclovir. Samples for PK assessments will be obtained to assess the exposure concentration. If the safety profile and the drug exposure concentrations in Cohort 1 are acceptable, eight new subjects will be enrolled in Cohort 2. The dose that these subjects will receive will be predicated upon the pharmacokinetic data from Cohort 1.

DETAILED DESCRIPTION:
A Phase 1, open label multicenter trial to assess the safety and pharmacokinetics (PKs) of oral valacyclovir in neonates who are at risk of acquiring neonatal herpes simplex virus disease. This study will determine the valacyclovir dose that results in a systemic acyclovir exposure comparable to 10 mg/kg of parenterally administered acyclovir, which is an AUC0-12 of 24,000 ngxhr/mL to 48,000 ngxhr/mL. Neonates whose mothers have a history of genital HSV infection and received oral valacyclovir in the last several weeks of pregnancy, as per the recommendations of the American College of Obstetrics and Gynecology (ACOG) (9), will be eligible for enrollment. Cohort 1 will be comprised of eight subjects. Following informed consent, each subject will receive 10 mg/kg of oral valacyclovir, and may start taking oral valacyclovir while still in the birth hospital, with subsequent dosing at home, or may start taking oral valacyclovir following discharge from the birth hospital. If the safety profile and the drug exposure concentrations in Cohort 1 are acceptable, eight new subjects will be enrolled in Cohort 2. The dose that these subjects will receive will be predicated upon the pharmacokinetic data from Cohort 1. The primary study objective is to establish the dose of valacyclovir in neonates that reliably achieves systemic acyclovir exposures comparable to 10 mg/kg of parenterally administered acyclovir. The secondary study objectives are: 1) to define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir and 2) to assess and describe the safety profile of valacyclovir among treated neonates.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s)
2. Maternal history of genital HSV infection
3. Maternal receipt of oral acyclovir, valacyclovir, or famciclovir suppressive therapy for >/= 7 days prior to delivery
4. Gestational age >/= 38 weeks at birth
5. </= 2 days of age at study enrollment*
6. Weight at study enrollment >/= 2,000 grams

   * For purposes of this study, the calendar day of birth is Day of Life 0

Exclusion Criteria:

1. Evidence of neonatal HSV infection
2. Evidence of sepsis
3. Known renal anomalies or dysfunction
4. Maternal genital lesions suspicious for HSV at the time of delivery
5. Infants known to be born to women who are HIV positive (but HIV testing is not required for study entry)
6. Current receipt in the neonate of acyclovir, ganciclovir, famciclovir, or any investigational drugs

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Neonatal plasma acyclovir mean AUC12 concentrations | Days 1 - 5
  To establish the dose of valacyclovir in neonates that reliably achieves systemic acyclovir exposures comparable to 10 mg/kg of parenterally administered acyclovir. Acyclovir target concentration of following oral valacyclovir dosing is 24,000 ngxhr/mL to 48,000 ngxhr/mL.

SECONDARY OUTCOMES:
Half-life (t1/2) of acyclovir | Days 1 - 5
  To define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir
Maximum Serum Concentration (Cmax) of acyclovir | Days 1 - 5
  To define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir
Occurrence of Grade 3 Adverse Events (AEs) | Days 1 - 42
  To assess and describe the safety profile of valacyclovir among treated neonates
Occurrence of Grade 4 Adverse Events and Serious Adverse Events | Days 1 - 42
  To assess and describe the safety profile of valacyclovir among treated neonates
Oral Clearance (CL/F) of acyclovir | Days 1 - 5
  To define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir
Time to the maximum concentration (Tmax) of acyclovir | Days 1 - 5
  To define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir
Volume of distribution (V/F) of acyclovir | Days 1 - 5
  To define the pharmacokinetic profile of acyclovir in neonates receiving oral valacyclovir

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Children's of Alabama Child Health Research Unit (CHRU), Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Louisville School of Medicine - Norton Children's Hospital - Infectious Diseases, Louisville, Kentucky
  - M Health Fairview Masonic Children's Hospital, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Children's Nebraska, Omaha, Nebraska
  - Steven and Alexandra Cohen Childrens Medical Center of New York - New Hyde Park - Infectious Disease, Queens, New York
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York
  - SUNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Atrium Health ID Consultants & Infusion Care Specialists, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin